CLINICAL TRIAL: NCT00395304
Title: Childhood Asthma Research and Education (CARE) Network Trial - Best Add-On Therapy Giving Effective Response (BADGER)
Acronym: BADGER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Vernon M. Chinchilli, PhD, Professor and Chair, Department of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 444; 5U10HL064313 (NIH); 5U10HL064288 (NIH); 5U10HL064305 (NIH); 5U10HL064295 (NIH); 5U10HL064287 (NIH); 5U10HL064307 (NIH)
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Results first posted 2010-09-17 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; montelukast; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Sequence #1 (Experimental): fluticasone propionate + montelukast, followed by fluticasone propionate, followed by fluticasone propionate + salmeterol
  Interventions: Drug: fluticasone propionate + montelukast; Drug: fluticasone propionate; Drug: fluticasone propionate + salmeterol
- Sequence #2 (Experimental): fluticasone propionate + montelukast, followed by fluticasone propionate + salmeterol, followed by followed by fluticasone propionate
  Interventions: Drug: fluticasone propionate + montelukast; Drug: fluticasone propionate; Drug: fluticasone propionate + salmeterol
- Sequence #3 (Experimental): fluticasone propionate + salmeterol, followed by fluticasone propionate, followed by fluticasone propionate + montelukast
  Interventions: Drug: fluticasone propionate + montelukast; Drug: fluticasone propionate; Drug: fluticasone propionate + salmeterol
- Sequence #4 (Experimental): fluticasone propionate + salmeterol, followed by fluticasone propionate + montelukast, followed by fluticasone propionate
  Interventions: Drug: fluticasone propionate + montelukast; Drug: fluticasone propionate; Drug: fluticasone propionate + salmeterol
- Sequence #5 (Experimental): fluticasone propionate, followed by fluticasone propionate + salmeterol, followed by fluticasone propionate + montelukast
  Interventions: Drug: fluticasone propionate + montelukast; Drug: fluticasone propionate; Drug: fluticasone propionate + salmeterol
- Sequence #6 (Experimental): fluticasone propionate, followed by fluticasone propionate + montelukast, followed by fluticasone propionate + salmeterol
  Interventions: Drug: fluticasone propionate + montelukast; Drug: fluticasone propionate; Drug: fluticasone propionate + salmeterol

INTERVENTIONS:
Drug: fluticasone propionate + montelukast — Dry-powder inhaler fluticasone 100 mcg bid (Flovent Diskus®, GlaxoSmithKline) plus Montelukast 5 or 10 mg qd (Singulair®, Merck)
  Other Names: Flovent Diskus® + Singulair®
Drug: fluticasone propionate — Dry-powder inhaler fluticasone 250 mcg bid (Flovent Diskus®, GlaxoSmithKline)
  Other Names: Flovent Diskus®
Drug: fluticasone propionate + salmeterol — Dry-powder inhaler fluticasone + salmeterol combination 100 mcg/50 mcg bid (Advair Diskus®, GlaxoSmithKline)
  Other Names: Advair Diskus®

SUMMARY:
Asthma is a common, serious illness among children in the United States. While a low dose of inhaled corticosteroids (ICS) may effectively control symptoms, some children may require additional medications to maintain adequate asthma control. This study compares the effectiveness of a higher dose of ICS, ICS combined with a long-acting beta-agonist (LABA) medication, and ICS combined with a leukotriene receptor antagonist (LTRA) medication at reducing the impact and severity of asthma exacerbations that occur in children with mild to moderate persistent asthma.

DETAILED DESCRIPTION:
Almost 9 million children in the United States have asthma, and it is a leading cause of hospitalizations and school absenteeism. Common asthma symptoms include wheezing, shortness of breath, chest tightness, and coughing. While there is no cure for asthma, most children who receive proper treatment are able to control symptoms and lead a normal life. Low doses of ICS are commonly prescribed to prevent symptoms and keep asthma under control. While this is usually sufficient to prevent asthma attacks, some children do not respond well to low dose ICS alone. For these children, their asthma symptoms may be more effectively controlled by either receiving a higher dose of ICS or receiving LABA or LTRA medications in combination with a low dose of ICS. Both LABA and LTRA medications are used to help control moderate to severe asthma. The purpose of this study is to compare the effectiveness of a high dose of ICS versus a low dose of ICS plus either LABA or LTRA medication at improving asthma control and reducing the severity of symptoms that occur in children with mild to moderate persistent asthma.

This study began with an 8-week screening period during which participants were monitored while they used an inhaler with a low dose of ICS medication. During this time, participants also attended one or two study visits. At each visit, participants underwent a physical examination, exhaled nitric oxide analysis, and lung function and airway pressure testing. After enrollment criteria were met, participants underwent these same evaluations again, and they completed questionnaires to assess asthma control, quality of life, and home environmental factors. Blood was collected and a methacholine challenge test was completed, which artificially triggers an asthma attack to determine the severity of an individual's asthma. Participants then were randomly assigned to one of six treatment sequences, each of which includes the following three regimens in a different order:

* Low dose of ICS and salmeterol, a LABA medication
* Low dose of ICS and montelukast, a LTRA medication
* Double dose of ICS

Each treatment period lasted 16 weeks, with study visits occurring weekly. A physical examination, blood collection, lung function and airway pressure testing, a methacholine challenge test, and questionnaires occurred at selected visits. Throughout the study, participants recorded asthma symptoms, peak expiratory flow rates, and rescue medication usage in a daily diary. The entire length of the study did not exceed 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to perform reproducible spirometry according to American Thoracic Society (ATS) criteria
* History of asthma symptoms (e.g., cough, wheezing, shortness of breath) and meets at least one of the following criteria:

  1. Naïve to controller therapy and meeting National Asthma Education and Prevention Program (NAEPP) criteria for mild-moderate persistent asthma (symptoms at least 2 days per week and/or night-time awakenings due to asthma at least 2 nights per month)
  2. Current uncontrolled asthma (meets NAEPP criteria for mild-moderate persistent asthma) while receiving an ICS dose greater than or equal to 200 ug per day of fluticasone equivalent or some form of non-ICS controller therapy (e.g., montelukast, theophylline, cromolyn)
  3. Asthma is currently under control while receiving an ICS dose between 300 to 400 ug per day of fluticasone equivalent and willing to consider changing current treatment to monotherapy with one dose of ICS (current standard of care)
  4. Asthma is currently under control while receiving some form of combination therapy, such as ICS less than or equal to 200 ug per day of fluticasone equivalent in addition to a non-ICS controller therapy (e.g., LABA, montelukast, theophylline, cromolyn), and willing to consider changing current treatment to monotherapy with one dose of ICS (current standard of care)
* FEV1 reversibility of at least 12% following bronchodilator administration (4 puffs) at study visit 1. Individuals will need to hold albuterol, montelukast, theophylline, ipratropium bromide (or other anticholinergics) and LABAs per study instructions prior to reversibility testing. If an individual is receiving these types of medications prior to study visit 1, he/she may be brought back to the clinical center within 1 week following appropriate medication withholding to attempt qualification by reversibility criteria. If the individual does not meet this requirement, they may qualify for enrollment if their PC20 methacholine FEV1 is less than or equal to 12.5 mg/ml at the time of randomization. If FEV1 is less than 70%, thus precluding the methacholine challenge at this visit, then completion of the visit will be postponed several days and an additional attempt to obtain a methacholine challenge test will be made. If the methacholine challenge still cannot be performed, an individual may still qualify by reversibility criteria at this visit.
* History of clinical varicella or varicella vaccine; individuals needing the vaccine may receive it from their primary care physician prior to study entry
* Ability of parent to provide informed consent; verbal assent must be obtained from children less than 7 years of age and written assent must be obtained from children between 7 and 18 years of age
* If female, willing to use an effective form of contraception

Prior to being randomly assigned to a treatment group, participants must meet the following criteria to remain in the study:

* Lack of acceptable asthma control during the 8-week screening period as defined by the following criteria:

  1) On average, on more than 2 days per week, one or all of the following:
  1. Diary-reported symptoms
  2. The use of inhaled bronchodilator (not including pre-exercise)
  3. Peak flows in the yellow zone (less than 80% of post bronchodilator PEF value obtained at study visit 1) OR
* On average, more than 1 night-time awakening due to asthma, during each 2-week period

Exclusion Criteria:

* Corticosteroid treatment for any condition prior to study entry within the following defined timepoints:

  1. Oral - Use within 2 weeks of the screening visit
  2. Injectable - Use within 2 weeks of the screening visit
  3. Nasal - May be used at any time during the study at the discretion of the study investigator or primary care physician
* Current or prior use of medications known to significantly interact with corticosteroid disposition (within a 2-week period of study visit 1), including but not limited to carbamazepine, erythromycin or other macrolide antibiotics, phenobarbital, phenytoin, rifampin, or ketoconazole
* Pre-bronchodilator FEV1 less than 60% predicted at study visit 1
* More than three hospitalizations for asthma in the year prior to study entry
* Presence of chronic or active lung disease other than asthma
* Significant medical illness other than asthma, including thyroid disease, diabetes mellitus, Cushing's disease, Addison's disease, hepatic disease, or concurrent medical problems that could require oral corticosteroids during the study or would place the participant at increased risk while participating in the study
* History of cataracts, glaucoma, or any other medical disorder associated with an adverse effect to corticosteroids
* Gastroesophageal reflux symptoms not controlled by standard medical therapy
* History of significant asthma exacerbation within 2 weeks of study visit 1 or more than 5 courses of systemic corticosteroids in the year prior to study entry
* History of a life-threatening asthma exacerbation requiring intubation, mechanical ventilation, or resulting in a hypoxic seizure within the 5 years prior to study entry
* History of adverse reactions to ICS, LTRA, or LABA preparations or any of their ingredients
* Receiving hyposensitization therapy other than an established maintenance regimen (i.e., continuous regimen for at least 3 months prior to study entry)
* Pregnant or breastfeeding
* Inability to perform study procedures
* Refusal to consent to a genotype evaluation
* Inability of the child to ingest the study drug
* Cigarette smoking or smokeless tobacco use in the year prior to study entry
* Current participation or participation in the month prior to study entry in another investigational drug trial
* Evidence that the family may be unreliable or nonadherent, or may move from the clinical center area before study completion

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2007-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T. Mauger, PhD, Principal Investigator — Penn State College of Medicine; Stanley J. Szefler, MD, PhD, Principal Investigator — National Jewish Health; Robert F. Lemanske, Jr., MD, Principal Investigator — University of Wisconsin, Madison; Robert S. Zeiger, MD, PhD, Principal Investigator — Kaiser Permanente Medical Center; Robert C. Strunk, MD, Principal Investigator — Washington University School of Medicine; Fernando D. Martinez, MD, Principal Investigator — University of Arizona College of Medicine; Lynn M. Taussig, MD, Study Chair — University of Denver
Locations (5):
- United States (5):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Kaiser Permanente Medical Center, San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin - Madison, Madison, Wisconsin

REFERENCES:
- [Result] Lemanske RF Jr, Mauger DT, Sorkness CA, Jackson DJ, Boehmer SJ, Martinez FD, Strunk RC, Szefler SJ, Zeiger RS, Bacharier LB, Covar RA, Guilbert TW, Larsen G, Morgan WJ, Moss MH, Spahn JD, Taussig LM; Childhood Asthma Research and Education (CARE) Network of the National Heart, Lung, and Blood Institute. Step-up therapy for children with uncontrolled asthma receiving inhaled corticosteroids. N Engl J Med. 2010 Mar 18;362(11):975-85. doi: 10.1056/NEJMoa1001278. Epub 2010 Mar 2. PMID 20197425
- See also: Click here for the Childhood Asthma Research and Education (CARE) Network web site — http://www.asthma-carenet.org

RESULTS

PARTICIPANT FLOW:
Groups:
- 2xICS, 1xICS + LABA, 1xICS + LTRA: Dry-powder inhaler fluticasone 250 mcg bid (Flovent Diskus®, GlaxoSmithKline), followed by Dry-powder inhaler fluticasone + salmeterol combination 100 mcg/50 mcg bid (Advair Diskus®, GlaxoSmithKline), followed by Dry-powder inhaler fluticasone 100 mcg bid (Flovent Diskus®, GlaxoSmithKline) plus Montelukast 5 or 10 mg qd (Singulair®, Merck)
- 2xICS, 1xICS + LTRA, 1xICS + LABA: Dry-powder inhaler fluticasone 250 mcg bid (Flovent Diskus®, GlaxoSmithKline), followed by Dry-powder inhaler fluticasone 100 mcg bid (Flovent Diskus®, GlaxoSmithKline) plus Montelukast 5 or 10 mg qd (Singulair®, Merck), followed by Dry-powder inhaler fluticasone + salmeterol combination 100 mcg/50 mcg bid (Advair Diskus®, GlaxoSmithKline)
- 1xICS +LABA, 2xICS, 1xICS + LTRA: Dry-powder inhaler fluticasone + salmeterol combination 100 mcg/50 mcg bid (Advair Diskus®, GlaxoSmithKline), followed by Dry-powder inhaler fluticasone 250 mcg bid (Flovent Diskus®, GlaxoSmithKline), followed by Dry-powder inhaler fluticasone 100 mcg bid (Flovent Diskus®, GlaxoSmithKline) plus Montelukast 5 or 10 mg qd (Singulair®, Merck)
- 1xICS + LABA, 1xICS + LTRA, 2xICS: Dry-powder inhaler fluticasone + salmeterol combination 100 mcg/50 mcg bid (Advair Diskus®, GlaxoSmithKline), followed by Dry-powder inhaler fluticasone 100 mcg bid (Flovent Diskus®, GlaxoSmithKline) plus Montelukast 5 or 10 mg qd (Singulair®, Merck), followed by Dry-powder inhaler fluticasone 250 mcg bid (Flovent Diskus®, GlaxoSmithKline)
- 1xICS + LTRA, 2xICS, 1xICS + LABA: Dry-powder inhaler fluticasone 100 mcg bid (Flovent Diskus®, GlaxoSmithKline) plus Montelukast 5 or 10 mg qd (Singulair®, Merck), followed by Dry-powder inhaler fluticasone 250 mcg bid (Flovent Diskus®, GlaxoSmithKline), followed by Dry-powder inhaler fluticasone + salmeterol combination 100 mcg/50 mcg bid (Advair Diskus®, GlaxoSmithKline)
- 1xICS + LTRA, 1xICS + LABA, 2xICS: Dry-powder inhaler fluticasone 100 mcg bid (Flovent Diskus®, GlaxoSmithKline) plus Montelukast 5 or 10 mg qd (Singulair®, Merck), followed by Dry-powder inhaler fluticasone + salmeterol combination 100 mcg/50 mcg bid (Advair Diskus®, GlaxoSmithKline), followed by Dry-powder inhaler fluticasone 250 mcg bid (Flovent Diskus®, GlaxoSmithKline)
Period: Treatment Period 1
Arm/Group | 2xICS, 1xICS + LABA, 1xICS + LTRA | 2xICS, 1xICS + LTRA, 1xICS + LABA | 1xICS +LABA, 2xICS, 1xICS + LTRA | 1xICS + LABA, 1xICS + LTRA, 2xICS | 1xICS + LTRA, 2xICS, 1xICS + LABA | 1xICS + LTRA, 1xICS + LABA, 2xICS
Started | 31 | 30 | 30 | 31 | 28 | 32
Completed | 30 | 26 | 30 | 28 | 27 | 30
Not Completed | 1 | 4 | 0 | 3 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | 2xICS, 1xICS + LABA, 1xICS + LTRA | 2xICS, 1xICS + LTRA, 1xICS + LABA | 1xICS +LABA, 2xICS, 1xICS + LTRA | 1xICS + LABA, 1xICS + LTRA, 2xICS | 1xICS + LTRA, 2xICS, 1xICS + LABA | 1xICS + LTRA, 1xICS + LABA, 2xICS
Started | 30 | 26 | 30 | 28 | 27 | 30
Completed | 30 | 22 | 29 | 27 | 27 | 28
Not Completed | 0 | 4 | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | 2xICS, 1xICS + LABA, 1xICS + LTRA | 2xICS, 1xICS + LTRA, 1xICS + LABA | 1xICS +LABA, 2xICS, 1xICS + LTRA | 1xICS + LABA, 1xICS + LTRA, 2xICS | 1xICS + LTRA, 2xICS, 1xICS + LABA | 1xICS + LTRA, 1xICS + LABA, 2xICS
Started | 30 | 22 | 29 | 27 | 27 | 28
Completed | 29 | 20 | 29 | 25 | 27 | 27
Not Completed | 1 | 2 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants randomized to the six crossover sequences
Arm/Group | All Participants
Number analyzed (Participants) | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 182
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 119
Region of Enrollment [Number; unit: participants]
  United States | 182

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a Differential Response to the Three Step-up Therapies Based on Fixed Threshold Criteria for the Following Three Asthma Control Measures: Use of Oral Prednisone for Acute Asthma Exacerbations, Asthma Control Days and FEV1.
Description: One treatment period was ranked as better than another if the total amount of prednisone received during the period was at least 180 mg less, if the number of annualized asthma-control days during the final 12 weeks of the period was increased by at least 31 days, or if the FEV1 at the end of the period was at least 5% higher. If the prednisone threshold was met, then we ignored the number of asthmacontrol days and the FEV1. If the threshold for asthma-control days was met, then we ignored the FEV1. Otherwise, the order of response was determined by the FEV1.
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: ITT. Although only 157 participants completed all three treatment periods, there was sufficient data on 8 additional participants to include them in the analysis of the primary outcome.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 165
Participants | 161

2. Secondary Outcome: Change From Baseline in the Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) % Predicted
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: Patients who completed the 16-week treatment period for the specific treatment (2xICS, 1xICS + LABA, or 1xICS + LTRA) within the three-way crossover design
Measure: Mean (Standard Deviation); unit: percentage points
Groups:
- 2xICS: Dry-powder inhaler fluticasone 250 mcg bid (Flovent Diskus®, GlaxoSmithKline)
- 1xICS + LABA: Dry-powder inhaler fluticasone + salmeterol combination 100 mcg/50 mcg bid (Advair Diskus®, GlaxoSmithKline)
- 1xICS + LTRA: Dry-powder inhaler fluticasone 100 mcg bid (Flovent Diskus®, GlaxoSmithKline) plus Montelukast 5 or 10 mg qd (Singulair®, Merck)
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 161 | 160 | 155
percentage points | 0.26 (11.02) | 1.07 (9.45) | -0.84 (10.25)

3. Secondary Outcome: Change From Baseline in the Post-bronchodilator FEV1 Percent Predicted
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 157 | 152 | 153
percentage points | -0.2 (9.7) | -1.2 (8.9) | -0.8 (10.1)

4. Secondary Outcome: Change From Baseline in the Pre-bronchodilator Forced Vital Capacity (FVC) % Predicted
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 161 | 160 | 155
percentage points | -1.00 (10.18) | -1.58 (8.04) | -1.56 (8.63)

5. Secondary Outcome: Change From Baseline in the Pre-bronchodilator FEV1/FVC Ratio
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 161 | 160 | 155
ratio | 0.98 (4.60) | 2.13 (4.75) | 0.55 (5.11)

6. Secondary Outcome: Change From Baseline in the Morning Peak Expiratory Flow Rate (PEFR) % Predicted
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 159 | 161 | 155
percentage points | 4.44 (11.25) | 6.26 (9.91) | 4.04 (9.66)

7. Secondary Outcome: Change From Baseline in the Evening Peak Expiratory Flow Rate (PEFR) % Predicted
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 159 | 161 | 155
percentage points | 2.84 (10.17) | 4.87 (9.20) | 2.29 (8.73)

8. Secondary Outcome: Change From Baseline in the Peak Expiratory Flow Rate (PEFR) Variability
Description: PEFR variability is calculated as 100% times the difference between the evening and morning PEFR values, divided by the average of the evening and morning PEFR values, i.e., PEFR variability = 100% x (morning PEFR - evening PEFR)/((morning PEFR + evening PEFR)/2)
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 154 | 156 | 150
percentage points | 2.09 (7.37) | 1.61 (6.83) | 1.72 (6.68)

9. Secondary Outcome: Change From Baseline in the Impulse Oscillometry Resistance at 5 Hertz
Description: Change from baseline in the impulse oscillometry resistance at 5 Hertz, measured in kiloPascals per liters per second
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kiloPascals per liters per second
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 165 | 163 | 161
kiloPascals per liters per second | -0.08 (0.15) | -0.09 (0.13) | -0.06 (0.14)

10. Secondary Outcome: Change From Baseline in the Logarithm Base 2 of the Methacholine PC20
Description: The methacholine PC20 is the concentration of methacholine that causes a 20% decrease in the pre-bronchodilator FEV1. The logarithm base 2 transformation converts the PC20 into doubling dilutions.
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: doubling dilutions
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 111 | 112 | 94
doubling dilutions | 1.11 (2.14) | 1.20 (2.31) | 1.00 (2.16)

11. Secondary Outcome: Change From Baseline in the Natural Logarithm of Exhaled Nitric Oxide (eNO)
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: natural logarithm of parts per billion
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 151 | 150 | 150
natural logarithm of parts per billion | -0.04 (0.68) | -0.05 (0.74) | -0.02 (0.71)

12. Secondary Outcome: Change From Baseline in the Asthma Control Test (ACT)
Description: The ACT consists of five items, each scored as 1 (worst) to 5 (best). The five items are averaged.
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 164 | 162 | 159
units on a scale | 1.49 (4.09) | 1.87 (4.12) | 1.69 (4.00)

13. Secondary Outcome: Change From Baseline in Asthma Quality of Life
Description: Asthma quality of life is measured as the average of 23 questions, each of which is scored from 1 (worse) to 7 (best)
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 165 | 161 | 160
units on a scale | 0.2 (0.1) | 0.3 (0.9) | 0.3 (1.0)

14. Secondary Outcome: Number of Participants With Asthma Exacerbations
Description: An asthma exacerbation was defined as the administration of a course of oral/systemic prednisone for the treatment of asthma.
Time Frame: Measured during the last 12 weeks of each 16-week treatment period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2xICS | 1xICS + LABA | 1xICS + LTRA
Number analyzed (Participants) | 165 | 163 | 161
Participants | 49 | 35 | 37

ADVERSE EVENTS:
Time Frame: 1 year
Description: does not differ from the clinicaltrials.gov definitions
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 7/182
Other Adverse Events (participants affected / at risk) | 22/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=182)
asthma exacerbation requirung hospitalization (Respiratory, thoracic and mediastinal disorders) | 3 (3)
appendicitis (Gastrointestinal disorders) | 1 (1)
tonsillectomy (Blood and lymphatic system disorders) | 2 (2)
behavioral problems (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=182)
asthma exacerbation not requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 22 (22)

LIMITATIONS AND CAVEATS:
The study was not designed or powered to evaluate the long-term safety of long-acting beta-agonists in children. The duration of the trial and its sample size preclude statements regarding long-term risks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No